CLINICAL TRIAL: NCT04762381
Title: Effect of 24 mg Dexamethasone Preoperatively on Surgical Stress, Pain and Recovery in Robotic-assisted Laparoscopic Hysterectomy
Brief Title: Dexamethasone and Robotic-assisted Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Collaborators: Hospital of Southern Jutland (Other)
Responsible Party: Principal Investigator, Finn Lauszus, Associate Professor, Hospital of Southern Jutland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Robotic surgery and steroid
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Response; Pain, Postoperative; Nausea, Postoperative; Incontinence; Sexual Behavior
Keywords: inflammatory response; surgical stress; leucocytes; IL-6; mRNA transcription; incontinence; sexual function; work life
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Sexual Behavior | interventions — dexamethasone 21-phosphate; Glucocorticoids

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded, results enteree into RedCap, logged and masked for participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): 24 mg dexamethasone as single dose intravenously peroperatively
  Interventions: Drug: Dexamethasone phosphate
- Placebo (Placebo Comparator): saline infusion intravenously in a single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone phosphate — 24 mg dexamethasone infused peroperatively
  Other Names: glucocorticoid
  Arms: Dexamethasone
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
Robotic-assisted hysterectomy is an alternative to laparoscopic surgery as part of a minimal invasive regimen. Several treatment strategies are followed to improve the overall outcome and minimize surgical stress. Glucocorticoids provide significant analgesic and antiemetic effects but its role in a fast-track, multi-modal setting is not settled when discharge is planned within 24-36 hours.

This study will evaluate in a randomized trial the effect of a single dose of 24 mg dexamethasone on women undergoing robotic-assisted hysterectomy with regard to surgical stress measured by c-reactive protein as primary outcome and, further, other stress markers like white blood cells. The postoperative recovery will be registered in validated charts and questionnaires for pain and analgesic use, quality of recovery, incontinence, sexual and work life. Furthermore, in a sub-analysis, transcriptional profiling will be applied to explore, which parts of the innate and cellular immune system is activated to explore the mechanisms of surgical stress response.

The hypothesis is that women undergoing robotic hysterectomy would benefit from peroperative glucocorticoid treatment on important life qualities like pain, fatigue, freedom of medications and resuming work and sexual activities. Further, future adjuvant peroperative regimens may be able to target the stress response in a more appropriate way

DETAILED DESCRIPTION:
Background Robotic operations in gynecology is one of the fastest growing fields in applied robotic technology.

In Denmark 4000 hysterectomies are performed each year on benign indications and minimal invasive techniques has risen from 35 to 80%. These operations consist of vaginal, laparoscopic assisted und the latest robotic assisted hysterectomy. Hysterectomy and prostate operations are the most common robotic assisted operations as an alternative to conventional laparoscopy.

Robotic surgery on benign indications in gynecology is still a discussion on the cost vs. benefit due to increased cost and lack of evidence on superiority in surgical outcome compared to conventional laparoscopy. For minimal invasive surgery is but a part of a complex series of treatment in a strategy, the so-called multi-modal regimen (1-7,16). By this, the day of discharge has dramatically decreased without compromising safety during surgery and postoperative recovery. However, not all single elements are proven for efficacy, let alone the specific targets for effect (16).

To further improve the overall outcome of surgery the surgical stress response are investigated, which includes inflammatory components and are of importance of postoperative pain and recovery (8,9,16). Here amongst others, glucocorticoids have proven to relieve pain in a number of procedures, applied in general surgery on colon, gallbladder, and breast, in orthopedic surgery on knee and breast surgery, and in gynecology, too, in laparoscopic hysterectomy (1-10,15,16). The dose of steroid to provide significant analgesic effect is, at least, dexamethasone of 0.1-0.2 mg/kg or 15 mg, which is substantiated in some reduction in inflammatory response (7,15,16). Glucocorticoids are known for analgesic, opioid-sparing and antiemetic effects but procedure-specific outcome are lacking. Similarly, the specific anti-inflammatory and sites of surgical stress-related responses are not well elucidated.

Aim The PhD study evaluate the effects of a single dose of steroid on acute postoperative stress response and pain after hysterectomy. The evaluation is on clinical relevant outcome that directly benefit the patients. We will measure surgical stress by c-reactive protein and other inflammatory markers based on transcriptional profiling, register pain and medication needed during hospital stay and after discharge, and when work and sexual function could be resumed.

Outcome The primary endpoint is reduction of postoperative c-reactive protein (crp) after robotic hysterectomy as an objective measurement of the stress amelioration by the given steroid. The rise postoperatively will be ascertained by two baseline measurements and every 4-6 hours after operation as long as the women is not discharged. The crp is not expected to be dependent on each operation team eagerness to perform well or the postoperative care to reach certain standards.

As secondary outcome we register pain scores from baseline to 24 h and later on, the postoperative analgesics medication from baseline to discharge and later on, quality of recovery (QoR-15D) in the latest 24 hours (12). Further, after discharge incontinence (ICIQ-UI), start of sexual life (PISQ-12/31), inflammatory markers, and resumption to recreational and work life will be ascertained in a diary. The baseline and early acute postoperative pain scores (visual analog scale, VAS) at rest and at movement (0-4 h postoperatively), late acute postoperative pain scores (VAS) at rest and at movement (24 h postoperatively); and cumulative opioid consumption (up to 24 h) will be registered. Part of blood samples will be stored for analysis of the cellular inflammatory systems by NanoString to explore the innate system and cellular activation (19,20). NanoString has the capacity to demonstrate activation of immune-related genes in the bloodstream during inflammatory induction and highlight an exciting role of immune competent cell in linking peripheral inflammation with immune activation and possibly anti-nociception. NanoString methodology investigates gene expression and currently quantifies the expression of 770 genes by determining the amount of messenger RNA (mRNA). mRNA is the end-product of gene transcription and, therefore, allows the study of gene up-regulation.

Monitoring cycles and levels of rest and activity will be done by an actigraph in a non-invasive method (13,14).

Hypothesis Women undergoing robotic hysterectomy would benefit from peroperative glucocorticoid treatment on important life qualities like pain, fatigue, freedom of medications and resuming work and sexual activities. Biological substrates such as inflammatory markers will be explored as underlying mechanism behind surgical stress response in order to direct perioperative medical interventions (19).

Perspectives and impact The randomized design will evaluate the effects of the single dose dexamethasone on the highest level of evidence. The anti-emetic effects of steroid are already incorporated in several guidelines on perioperative care; however, this study could further enhance our knowledge on minimal invasive surgery and optimize the treatment for surgical stress. The stress response in humans have evolved over millennia and is embedded in our genes but has no natural association with modern days surgery and may be ill placed and timely inadequate for recovery. The exploratory study may help identify pathways and specific mechanism in surgical stress that can be targeted in future to enhance women's recovery after surgery. The perspective is in further studies to target these specific sites in the immune activation.

Methods:

The PhD study in robotic hysterectomy will include a randomized trial with a single dose intravenously of 24 mg dexamethasone (Dexavit®) corresponding to 128 mg methyl prednisolone (Solumedrol®).

The randomization will be performed in Redcap and data stored the same place under each patient cpr.-no. but in a separate section. A person not involved in the project in any other form will perform the randomization. The patient will then receive the dose of either steroid or placebo saline intravenously, blinded to the patient and operation team (gynecology, operation ward and anesthesiology). The applicant PhD student will later enter the data in Redcap unknowing to the randomization results.

All women in the department operated by with a robotic assisted hysterectomy will be monitored and fill out a diary with validated questionnaires (names of quest.) to streamline the information gathering in a high flow work place and not to discriminate those outside of the project. These data will be presented as the drop-out analysis to evaluate the external validity of the trial. The flow of data collection is displayed below.

Sample size was calculated to be 49 women included in each arm on the primary outcome of c-reactive protein rising to the level of 40 mg/l with an expected reduction of 10 % a with a standard deviation of 7 calculated by https://clincalc.com/stats/samplesize.aspx (1,17,18). This may seem a parsimonious reduction but in practical terms, it translates to more than halving the need of opioids early and late postoperatively (2). On the assumption of incomplete data in less than 10 % of cases, 50 women in each group with complete data will be included. Robotic hysterectomy is a standard procedure in our department with about 80-90 hysterectomies each year, so we expect the study inclusion to last 1½-2 years.

Statistics Analysis are performed on the intention-to-treat principle with women on current use of analgesics as a subgroup analysis. The statistics will be unpaired and paired analysis (2-ways ANOVA) including relevant co-variates. Regression analysis will be performed with the primary outcome as dependent variable and the secondary outcomes and anthropometrics as dependent variable.

ELIGIBILITY:
Inclusion Criteria:

* Meno-metrorrhagia,
* dysmenorrhea,
* fibroma,
* dysplasia,
* dysmenorrhea,
* ability in Danish writing

Exclusion Criteria:

* current treatment with glucocorticoids, opioids and NSAID analgesics,
* diabetes,
* current treatment of malignant disease,
* renal or hepatic disease,
* unable to communicate in Danish language.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
level of c-reactive protein (CRP) | 0-36 hours
  c-reactive protein measured in mg/l

SECONDARY OUTCOMES:
level of IL-6 | 0-36 hours
  Interleukin 6
Leucucytes | 0-36 hours
  White blood cell count
mRNA | 0-36 hours
  Transcription of mRNA after surgery
Incontinence | 0-14 days
  ICIQ-UI postoperatively
Sexual function | 0-14 days
  PISQ-12 postoperatively
work life checklist | 0-14 days
  Diary postoperatively
Number of steps count measured by pedometer | 0-14 days
  daily activity

CONTACTS AND LOCATIONS:
Overall Officials: Britta Frederiksen, PhD, Study Chair — Gyn. Dept. Aabenraa Hospital, Sygehus Sønderjylland
Locations (1):
- Gyn. Dept.;Aabenraa Hospital, Sygehus Sønderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: Yes
after PhD submission and evaluation and publiaction of results the data can be shared anonymously
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2025
Access Criteria: personal contact

REFERENCES:
- [Background] Lunn TH, Kristensen BB, Andersen LO, Husted H, Otte KS, Gaarn-Larsen L, Kehlet H. Effect of high-dose preoperative methylprednisolone on pain and recovery after total knee arthroplasty: a randomized, placebo-controlled trial. Br J Anaesth. 2011 Feb;106(2):230-8. doi: 10.1093/bja/aeq333. Epub 2010 Dec 3. PMID 21131371
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Jokela RM, Ahonen JV, Tallgren MK, Marjakangas PC, Korttila KT. The effective analgesic dose of dexamethasone after laparoscopic hysterectomy. Anesth Analg. 2009 Aug;109(2):607-15. doi: 10.1213/ane.0b013e3181ac0f5c. PMID 19608838
- [Background] Steinthorsdottir KJ, Kehlet H, Aasvang EK. Surgical stress response and the potential role of preoperative glucocorticoids on post-anesthesia care unit recovery. Minerva Anestesiol. 2017 Dec;83(12):1324-1331. doi: 10.23736/S0375-9393.17.11878-X. Epub 2017 Jun 12. PMID 28607335
- [Background] Lirk P, Thiry J, Bonnet MP, Joshi GP, Bonnet F; PROSPECT Working Group. Pain management after laparoscopic hysterectomy: systematic review of literature and PROSPECT recommendations. Reg Anesth Pain Med. 2019 Apr;44(4):425-436. doi: 10.1136/rapm-2018-100024. Epub 2019 Feb 3. PMID 30914471
- [Background] Wijk L, Nilsson K, Ljungqvist O. Metabolic and inflammatory responses and subsequent recovery in robotic versus abdominal hysterectomy: A randomised controlled study. Clin Nutr. 2018 Feb;37(1):99-106. doi: 10.1016/j.clnu.2016.12.015. Epub 2016 Dec 23. PMID 28043722